CLINICAL TRIAL: NCT05389436
Title: Comparison Between Outpatient and Inpatient Surgically Treated Ankle Fractures
Brief Title: Outpatient Versus Inpatient Surgery for Ankle Fractures
Acronym: OVISAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Grundtvig Refstrup Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Christian Grundtvig Refstrup Rasmussen, Principle investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20220012
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Ankle Fractures; Orthopedic Procedures; Surgical Procedures; Inpatient
MeSH Terms: conditions — Ankle Fractures | interventions — Ambulatory Care; Hospitalization

STUDY DESIGN:
Intervention Model Description: This study is a single center, prospective, assessor-blinded, randomized independent clinical trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of this study the patient, surgeon and care providers can not be blinded. The outcome assessor will be blinded with regards to the two treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The patient is discharged from the ER following X-ray, casting, charts. The patient is contacted when surgery is scheduled, and this is performed in a ambulatory setting
  Interventions: Procedure: Ambulatory care
- Standard (Active Comparator): The patient is admitted from the ER, surgery is performed when possible in regards to surgical capacity and swelling. Discharged when mobilised with cast.
  Interventions: Procedure: Inpatient care

INTERVENTIONS:
Procedure: Ambulatory care — The surgery is performed in ambulatory setting
  Arms: Experimental
Procedure: Inpatient care — The surgery is performed during inpatient care
  Arms: Standard

SUMMARY:
This study is a single center randomized controlled trail in which we compare outpatient and inpatient patients with an ankle fracture requiring surgical treatment.

DETAILED DESCRIPTION:
This study is a single center randomized controlled trail in which we compare outpatient and inpatient patients with an ankle fracture requiring surgical treatment.

Primary outcome: The primary objective of this study is to compare the 12-weeks patient reported Foot and Ankle Outcome Score (FOAS).

Secondary outcomes: Multiple other analysis are planned, but being secondary, they are hypothesis generating. They will include, but are not limited to, cross-over, unscheduled contacts, adverse events, pain, general health, time to return to work and socio-economic consequences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Ankle fracture indicating surgical treatment.
* Fracture stable in lower leg cast.
* Patient 18 years or older.
* Patient is able to ambulate with walking aid, and perform ADL at home.

Exclusion Criteria:

* Impaired physical, mental or social capacity incapable of participating in study.
* Incapable of reading or understanding Danish.
* Patient does not wich to participate.
* Concurrent major fracture to lower extremity (ipsi- and/or contralateral)
* Patholocigal fracture
* ASA score 3 or higher.
* Pregnancy.
* Open fracture.
* Infectious disease requiring isolation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Outcomes Score | 12 weeks
  The FAOS is a patient-reported structure-specific questionnaire. Consisting of 5 subscales: pain, symptoms, activities of daily living (ADL), function in sport and recreation (Sport/Rec), and foot- and ankle-related quality of life (QOL). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The result can be plotted as an outcome profile.

SECONDARY OUTCOMES:
Patient satisfaction | 2, 6 and 12 weeks
  Patient reported satisfaction. The patient is asked:
  1. "Given your experience with the treatment, how likely is it that you would choose it again?" and the possible answers are preplanned, using a 5 point Lickert scale: Very likely, likely, either/or, unlikely, very unlikely.
  2. "Given your experience with the treatment, how likely is it, that you would recommend it to a relative or friend?" and the possible answers are preplanned, using a 5 point Lickert scale: Very likely, likely, either/or, unlikely, very unlikely.
EQ-5D-5L questionnaire (5-level version) | 2, 6 and 12 weeks
  General health will be assessed using EQ-5D-5L questionnaire (5-level version), both the descriptive index and the EQ-VAS. It consists of five dimensions: Mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a self-rated health scale on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. An Eq5d-5L index of 1.0 indicated full health, 0 death, and -0.59 denoted a condition worse than death.
Tegner activity scale | 12 weeks
  The Tegner activity scale is a 1-item instrument that assesses activity levels for sports (competitive or recreational) and occupational activities (light or heavy labor). It evaluates the patient's level of work and sports activity on an 11-level scale, with higher scores representing higher levels of physical activity.
Adverse events | 2 days, 2, 6 and 12 weeks
  Adverse events, defined as any negative or unwanted reactions to the two groups will be recorded. Based on previous reports we will focus on: infection, DVT and re-operation. Patients are continuously requested to report any suspicion of a potential AE. Patients will be asked about potential AEs. Furthermore, medical records will be checked at the primary endpoint (12 weeks) for all AEs occurring from inclusion until the 12 week follow-up. An AE is defined as any undesirable experience during follow-up leading to contact with the healthcare system (general practitioner or hospital). If an AE result in hospitalization, prolonged inpatient hospital care, result in re-surgery, or if an AE is life-threatening, result in death, permanent disability or damage, they will be categorized as serious adverse events (SAEs).
Time to return to work | 2, 6 and 12 weeks
  The time from surgery to end of sick leave measured in days.
Bone union | 6 and 12 weeks
  Bone union, will be evaluated on standard AP and side X-rays of the fractured ankle. The evaluation of bone union will be defined as: i) visible callus formation, diminished no visible fracture line and no pain from the fracture site at weight-bearing and at clinical examination.
Pain intensity measured on a 10 cm VAS scale | 2 days, 2, 6 and 12 weeks
  Development in pain will be recorded by patient-reported pain intensity measured on a 10 cm visual analogue scale (VAS) with endpoints "no pain" and "maximal pain" for the worst pain during the last 24 hours and resting pain.
Ankle range of motion | 6 and 12 weeks
  Ankle range of motion. With the patient supine on an examination table the full range of passive motion in both ankle joints will be measured using a standard goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Christian GR Rasmussen, MD, Principal Investigator — Department of Orthopedic Surgery
Locations (1):
- Aalborg Universitetshospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No
A detailed statistical analysis plan will be made publicly available before the last patient is included in the study.

REFERENCES:
- [Derived] Rasmussen CG, Larsen P, Pedersen C, Elsoe R. Outpatient versus inpatient surgery for ankle fractures - a protocol for a randomised controlled trial. Dan Med J. 2025 Jun 26;72(7):A10240746. doi: 10.61409/A10240746. PMID 40600684